CLINICAL TRIAL: NCT06845852
Title: A Phase 1, Open-Label Study to Assess the Absorption, Metabolism, Excretion, and Mass Balance of [14C]Varegacestat Following a Single Oral Dose in Healthy Adult Male Participants
Brief Title: A Phase 1 Mass Balance Study of Varegacestat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immunome, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AL102-504
Record Dates: First submitted 2025-02-05; First posted 2025-02-25 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer
Keywords: absorption; metabolism; excretion; mass balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Drug: varegacestat (Experimental): Single oral dose of varegacestat administered on study Day 1
  Interventions: Drug: varegacestat

INTERVENTIONS:
Drug: varegacestat — Single oral dose of varegacestat

SUMMARY:
This clinical study is designed to study the mass balance of a single dose of varegacestat in healthy male participants.

DETAILED DESCRIPTION:
This is a single-center, open-label, Phase 1, mass balance study of varegacestat administered as a single oral dose (containing ~100 µCi) [14C]varegacestat in 6 healthy male participants.

Following completion of Screening and Day -1 assessments and an overnight fast of at least 10 hours, eligible participants will be administered a single dose (containing ~100 µCi) [14C]varegacestat as 2 oral capsules followed by approximately 240 mL room temperature filtered water on the morning of Day 1. Whole blood, plasma, urine, feces, and vomitus (if any, up to 24 hours post-dose) will be collected over at least 168 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Be a male participant between 18 and 55 years of age, inclusive, at Screening.
* Medically healthy based on the absence of clinically significant abnormal vital sign measurements, clinical laboratory test results (especially tests for renal and hepatic function), resting 12-lead Electrocardiogram (ECG) evaluation, and physical examination, as determined by the Investigator at Screening and the Check-In visit.

Exclusion Criteria:

* Have taken an investigational drug or participated in a clinical trial evaluating an investigational drug or device within 30 days (or 5 half-lives) prior to the study drug dose, whichever is longer.
* Have participated in a radiolabeled drug study or have been otherwise exposed to significant diagnostic (excluding dental X-rays), therapeutic, or occupational radiation, where exposure is made known to the Investigator, within one year prior to admission to the clinic for this study. The total estimated 12-month exposure to radio material or ionizing radiation should be below the CFR recommended levels considered safe (per US Title 21 CFR 361.1) or below 3000 mrem.
* Any condition which, in the opinion of the Investigator and/or Sponsor, would jeopardize participant safety or compliance with the Protocol.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
The mass balance of varegacestat following administration of a single oral dose (containing ~100 µCi) [14C]varegacestat in healthy adult male participants. | Up to 15 days

SECONDARY OUTCOMES:
The total radioactivity in plasma, whole blood, urine, and feces following administration of a single oral dose (containing ~100 µCi) [14C]varegacestat in healthy adult male participants. | Up to 15 days
The area under the concentration equivalent-time curve (AUC), from time 0 to the last observed non-zero concentration of varegacesatat and AL102-MTB (Varegacestat metabolite) in plasma. | Up to 15 days
The AUC from time 0 extrapolated to infinity, calculated as the sum of AUC0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant of varegacesatat and AL102-MTB in plasma. | Up to 15 days
Maximum observed concentration (Cmax) of varegacesatat and AL102-MTB (Varegacestat metabolite) in plasma. | Up to 15 days
Apparent first-order terminal elimination half-life (t1/2) will be calculated as 0.693/Kel of varegacesatat and AL102-MTB (Varegacestat metabolite) in plasma. | Up to 15 days
Percentage of each metabolite in urine and feces relative to the administered dose or percentage of metabolites in plasma relative to total drug related exposure AUC. | Up to 15 days
The safety and tolerability of a single oral dose (containing ~100 µCi) [14C]varegacestat in healthy adult male participants by incidences of treatment-emergent adverse events. | Up to 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Frontage Laboratories, Inc., Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided